CLINICAL TRIAL: NCT01796327
Title: A Phase 1, Single Dose, Fixed Sequence Study To Estimate The Absolute Bioavailability Of Dacomitinib (PF-00299804) By Comparing Oral To Intravenous Administration In Healthy Volunteers
Brief Title: A Study To Assess Absorption Of Study Drug Dacomitinib (PF-00299804), Given As An Oral Tablet Compared To An Intravenous Infusion In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A7471046
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: dacomitinib; PF-00299804; pharmacokinetics; bioavailability
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Dacomitinib will be administered as a single oral dose and as an intravenous infusion
  Interventions: Drug: dacomitinib oral; Drug: dacomitinib intravenous

INTERVENTIONS:
Drug: dacomitinib oral — Dacomitinib 45 mg oral tablet
Drug: dacomitinib intravenous — Dacomitinib 20 mg solution will be given as 1 hour intravenous infusion

SUMMARY:
This study aims to determine the proportion of study drug dacomitinib or PF-00299804, that is taken up from the digestive tract into the body when given as an oral tablet compared with that taken up by an intravenous dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female (of non-childbearing potential) subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Treatment with an investigational drug within 3 months or 5 half-lives preceding the first dose of study medication, whichever is longer.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Any known allergies or sensitivity to drug excipients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dacomitinib Dose-normalized Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. normalized to the administered dose
Dacomitinib Dose-normalized Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. normalized to the administered dose

SECONDARY OUTCOMES:
Dacomitinib Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Dacomitinib Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Dacomitinib Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t) normalized to the administered dose
Dacomitinib Maximum Observed Plasma Concentration (Cmax) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
Dacomitinib Time to Reach Maximum Observed Plasma Concentration (Tmax) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
Dacomitinib Apparent Oral Clearance (CL/F) | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Dacomitinib Apparent Volume of Distribution (Vz/F) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
PF-05199265 Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose
PF-05199265 Dose-normalized Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following oral dose normalized by administered dose
PF-05199265 Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
PF-05199265 Dose-Normalized Area Under the Curve From Time Zero to Last PF-05199265 Quantifiable Concentration [AUC (0-t)] following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t) normalized to the administered dose
Plasma Decay Half-Life (t1/2) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
PF-05199265 Maximum Observed Plasma Concentration (Cmax) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
Dacomitinib Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose
Dacomitinib Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Dacomitinib Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t) normalized to the administered dose
Dacomitinib Maximum Observed Plasma Concentration (Cmax) following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
Plasma Decay Half-Life (t1/2) of dacomitinib following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Systemic Clearance (CL) of dacomitinib following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution at Steady State (Vss) of dacomitinib following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
PF-05199265 Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose
PF-05199265 Dose-normalized Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  Area under the Concentration-Time Curve (AUC) From Time Zero to Extrapolated Infinite Time following intravenous dose normalized by administered dose
PF-05199265 Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
PF-05199265 Dose-Normalized Area Under the Curve From Time Zero to Last PF-05199265 Quantifiable Concentration [AUC (0-t)] following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t) normalized to the administered dose
PF-05199265 Maximum Observed Plasma Concentration (Cmax) following intravenous dose | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
Metabolite ratio for AUCinf after oral administration | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of AUCinf
Metabolite ratio for AUClast after oral administration | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of AUClast
Metabolite ratio for Cmax after oral administration | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of Cmax
Metabolite ratio for AUCinf after intravenous administration | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of AUCinf
Metabolite ratio for AUClast after intravenous administration | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of AUClast
Metabolite ratio for Cmax after intravenous administration | 0, 0.5, 1, 1.083, 1.25, 1.5, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  PF-05199265/dacomitinib ratio of Cmax
PF-05199265 Time to Reach Maximum Observed Plasma Concentration (Tmax) following oral dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
PF-05199265 Time to Reach Maximum Observed Plasma Concentration (Tmax) following IV dose | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ruddington Fields, Nottingham, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471046